CLINICAL TRIAL: NCT01723670
Title: A Double-Blind, Randomized, Placebo-Controlled, Multicenter Study to Evaluate the Effects of Multiple Dose Regimens of CHF 5074 for up to 2 Years on Potential Biomarkers of Neurodegeneration in Subjects With Mild Cognitive Impairment
Brief Title: Evaluation of Effects of Multiple Dose Regimens of CHF 5074 on Potential Biomarkers of Neurodegeneration in Subjects With Mild Cognitive Impairment
Acronym: CT05
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: CERESPIR (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CCD-1109-PR-0072
Record Dates: First submitted 2012-10-31; First posted 2012-11-08 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CHF 5074 1x (Experimental): oral tablet, multidose
  Interventions: Drug: CHF 5074 1x
- CHF 5074 2x (Experimental): oral tablet, multidose
  Interventions: Drug: CHF 5074 2x
- Placebo (Placebo Comparator): placebo, oral tablet, multidose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CHF 5074 1x — oral tablet, 1x, once a day for 24 months
  Arms: CHF 5074 1x
Drug: CHF 5074 2x — oral tablet, 2x, once a day for 24 months
  Arms: CHF 5074 2x
Drug: Placebo — oral tablet,once a day for 24 months
  Arms: Placebo

SUMMARY:
To evaluate the effects of multiple dose regimens of CHF 5074 administered once per day up to 2 years on potential biomarkers of neurodegeneration in subjects with mild cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* One or two Ɛ4 alleles of the apolipoprotein E (APOE) gene.
* Diagnosis of amnestic Mild Cognitive Impairment.
* Mini-Mental State Examination score higher than 24 at screening.

Exclusion Criteria:

* Diagnosis of Alzheimer's disease.
* Any medical condition that could explain the subject's cognitive deficits.
* MRI scans having evidence of pre-specified brain abnormalities.
* History of stroke.
* Vitamin B12 or folate deficiency.
* Skin cancers and any cancer that is being actively treated.
* Diagnosis of schizophrenia or recurrent mood disorder.
* Abnormal kidney function.
* Concomitant use of any study prohibitive medication.

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
To determine the effects on change from baseline on brain atrophy | pre-dose, Months 6, 12, 18, 24 and Washout

SECONDARY OUTCOMES:
To determine the presence of other biomarkers of neuronal degeneration | Day 1
To determine the presence of other biomarkers of neuronal degeneration | Month 24

OTHER OUTCOMES:
Change from baseline in cognitive performance | pre-dose, Month 6, Month 12, Month18, Month 24
  rate of cognitive decline
Change from baseline in global clinical status | pre-dose, Month 6, Month 12, Month 18, Month 24

CONTACTS AND LOCATIONS:
Overall Officials: Joel S Ross, MD, Principal Investigator — Memory Enhancement Center of America